CLINICAL TRIAL: NCT00450814
Title: Phase I/II Trial of Systemic Administration of Edmonston Strain of Measles Virus, Genetically Engineered to Express NIS, With or Without Cyclophosphamide, in Patients With Recurrent or Refractory Multiple Myeloma
Brief Title: Vaccine Therapy With or Without Cyclophosphamide in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC038C; NCI-2009-01194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC038C (Other: Mayo Clinic); P30CA015083 (NIH); R01CA125614 (NIH); R01CA168719 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 (MV-NIS alone) (Experimental): Patients receive MV-NIS IV over 1 hour on day 1. (Closed to accrual on 12/17/2009 and reopened 10/13/2011)
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter; Other: Pharmacological Study
- Stage 2 (MV-NIS and cyclophosphamide) (Experimental): Patients receive cyclophosphamide IV over 30 minutes and then MV-NIS IV over 1 hour 2 days later. (Temporarily closed to accrual on 10/13/11)
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Stage 2 (MV-NIS and cyclophosphamide)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter — Given IV
  Other Names: MV-NIS
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of vaccine therapy when given with or without cyclophosphamide and to see how well they work in treating patients with multiple myeloma that has come back (recurrent) or has not responded to previous treatment (refractory). Vaccines made from a gene-modified virus may help the body build an effective immune response to kill cancer cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving vaccine therapy together with cyclophosphamide may be a better treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) when administered with or without cyclophosphamide in patients with relapsed or refractory multiple myeloma. (Phase I) II. To evaluate the confirmed response rate of MV-NIS alone in patients with relapsed or refractory multiple myeloma who have exhausted all therapeutic options. (Phase II, Cohort A) III. To evaluate the confirmed response rate of MV-NIS alone in patients who are relapsing from very good partial response (VGPR) or complete response (CR) and have not received myeloma directed therapy for at least 12 weeks. (Phase II, Cohort B)

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity of the intravenous administration of an Edmonston vaccine strain measles virus engineered to express the thyroidal sodium iodide symporter (MV-NIS) when administered with or without cyclophosphamide in patients with relapsed or refractory multiple myeloma. (Phase I) II. To evaluate the confirmed response rate of MV-NIS in patients with relapsed or refractory multiple myeloma. (Phase I) III. To further evaluate the adverse event profile of MV-NIS in patients with relapsed or refractory multiple myeloma. (Phase II) IV. To evaluate overall survival, failure-free survival and progression-free survival. (Phase II)

TERTIARY OBJECTIVES:

I. To determine the time course of viral gene expression and virus elimination, and the biodistribution of virally infected cells at various times points after infection with MV-NIS (when administered with or without cyclophosphamide) using 99m-technetium (Tc) gamma camera imaging. (Phase I and II) II. To assess virus replication, viremia, viral shedding in urine and respiratory secretions, and virus persistence after systemic administration of MV-NIS (when administered with or without cyclophosphamide). (Phase I and II) III. To monitor humoral responses to the injected virus. (Phase I and II) IV. To explore the anti-myeloma efficacy (i.e. clinical response rate, time to progression, progression free survival, duration of response) of the virus using standard myeloma response criteria as well as immunoglobulin free light chain measurements. (Phase I and II)

OUTLINE: This is a phase I, dose-escalation study of MV-NIS followed by a phase II study. Patients are assigned to 1 of 2 treatment arms (Stage 1 or Stage 2) in phase I and assigned to Stage 1 in phase II.

STAGE 1 (MV-NIS ALONE, closed to accrual on 12/17/2009 and reopened 10/13/2011): Patients receive MV-NIS intravenously (IV) over 1 hour on day 1.

STAGE 2 (MV-NIS AND CYCLOPHOSPHAMIDE, temporarily closed to accrual on 10/13/11): Patients receive cyclophosphamide IV over 30 minutes and then MV-NIS IV over 1 hour 2 days later.

After completion of study treatment, patients are followed up at 6 weeks, 12 weeks, and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma relapsing from partial response or better

  * Patients relapsing > 18 months from transplant if not on maintenance, or
  * If off maintenance, discontinued at least 6 months ago, or
  * If relapsing on maintenance, at least 3 years from transplant, or
  * Off prior myeloma therapy at least 6 months ago
  * Sufficient tumor burden that is assessable for response

    * Serum M-spike >= 0.5 g/dL, or
    * If immunoglobulin A (IgA) myeloma, IgA > 1000 mg/dL, or
    * Difference between involved and uninvolved free light chain (dFLC) > 10 mg/dL, or
    * Urine M-spike >= 200 mg/24 hours, or
    * Bone marrow plasmacytosis >= 10%, or
    * Plasmacytoma >= 2 cm in diameter
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets (PLT) >= 50,000/uL
* Hemoglobin >= 8.5 g/dl
* Aspartate aminotransferase (AST) =< 2 times upper limit of normal
* Creatinine < 2 times upper limit of normal
* Total bilirubin =< 1.5 x upper limit of normal
* International normalized ratio (INR) =< 1.4 x ULN at the time of registration
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Willingness to provide all biological specimens as required by the protocol
* Negative serum pregnancy test done =< 7 days prior to registration for women of childbearing potential only
* Measles antibody titer on the BioRad Multiplex assay less than or equal to 1.0

Exclusion Criteria:

* Uncontrolled infection
* Active tuberculosis
* Any myeloma directed therapy within 12 weeks of registration including plasmapheresis or transfusion
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review
* Active central nervous system (CNS) disorder or seizure disorder
* Human immunodeficiency virus (HIV) positive test result
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (used for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation)
* Previous exposure to heat inactivated measles virus vaccine (this vaccine was given to some individuals between the years of 1963-1967)
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* Evidence of chronic or acute graft versus host disease or on-going treatment for graft versus host disease from prior allogeneic stem cell transplantation
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11-30 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I: INITIALLY CLOSED ON 12/17/2009 AND STAGE 2 BEGUN; HOWEVER, DUE TO NEW MANUFACTURING CAPABILITIES, STAGE 1 RE-OPENED ON October 13, 2011, FOR DOSE LEVELS 5 AND 6. Phase II: Accrual to Cohort A closed due to failed interim analysis. Cohort B closed due to lack of accrual.
Groups:
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 1: Patients receive 1x10^6 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 2: Patients receive 1x10^7 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 3: Patients receive 1x10^8 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 4: Patients receive 1x10^9 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 5: Patients receive 1x10^10 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 1 (MV-NIS Alone) Dose Level 6: Patients receive 1x10^11 MV-NIS (TCID50) IV over 1 hour on day 1.
- Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1: Patients receive 10 mg/kg cyclophosphamide IV over 30 minutes and then (Stage 1 MTD/100=10^7) MV-NIS (TCID50) IV over 1 hour 2 days later. (Temporarily closed to accrual on 10/13/11)
- Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2: Patients receive 10 mg/kg cyclophosphamide IV over 30 minutes and then 3 x 10^7 MV-NIS (TCID50) IV over 1 hour 2 days later. (Temporarily closed to accrual on 10/13/11)
- Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3: Patients receive 10 mg/kg cyclophosphamide IV over 30 minutes and then 9 x 10^7 MV-NIS (TCID50) IV over 1 hour 2 days later. (Temporarily closed to accrual on 10/13/11)
- Phase II (Acetaminophen + Benadryl + MV-NIS) Cohort A: Cohort A patients (relapsed or refractory multiple myeloma who have exhausted all therapeutic options) receive 650 mg Acetaminophen and 50 mg Benadryl orally 30 minutes prior to MV-NIS then receive MV-NIS IV over 1 hour on day 1.
- Phase II (Acetaminophen + Benadryl + MV-NIS) Cohort B: Cohort B patients (relapsing from VGPR or CR and have not
  > received myeloma directed therapy for at least 12 weeks) receive 650 mg Acetaminophen and 50 mg Benadryl orally 30 minutes prior to MV-NIS then receive MV-NIS IV over 1 hour on day 1.
Period: Overall Study
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3 | Phase II (Acetaminophen + Benadryl + MV-NIS) Cohort A | Phase II (Acetaminophen + Benadryl + MV-NIS) Cohort B
Started | 3 | 3 | 3 | 4 | 4 | 7 | 3 | 3 | 2 | 12 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 2 | 11 | 4
Not Completed | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Failed to complete the initial therapy | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Patient withdrawal prior to treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating early in Cohort B.
Groups:
- Phase II (Acetaminophen + Benadryl + MV-NIS): Patients receive 650 mg Acetaminophen and 50 mg Benadryl orally 30 minutes prior to MV-NIS then receive MV-NIS IV over 1 hour on day 1.
- Total: Total of all reporting groups
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3 | Phase II (Acetaminophen + Benadryl + MV-NIS) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 2 | 15 | 44
Age, Continuous [Median (Full Range); unit: years] | 64 [59 to 66] | 66 [57 to 68] | 51 [43 to 74] | 65 [63 to 82] | 63 [56 to 65] | 59 [49 to 65] | 62 [49 to 81] | 60 [59 to 65] | 65 [59 to 71] | 59 [40 to 72] | 60 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 1 | 5 | 1 | 1 | 0 | 4 | 18
  Male | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 2 | 2 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 2 | 13 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 0 | 0 | 1 | 0 | 3 | 5 | 2 | 2 | 1 | 9 | 23
    1 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 5 | 15
    2 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Participants With Dose-Limiting Toxicity Events (Phase I)
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Dose-limiting toxicities include non-hematologic events graded 3 or higher and deemed at least possibly related to treatment. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. The number of patients reporting a dose-limiting event are reported.
Time Frame: 6 weeks
Population: Only phase I patients who completed the study are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Dose-limiting toxicities include non-hematologic events graded 3 or higher and deemed at least possibly related to treatment. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. The MTD is reported below.
Time Frame: 6 weeks
Population: Only phase I stage 1 patients who completed the study are included in this analysis. Dose levels 1-6 of Phase I Stage 1 patients were combined in this analysis to determine the MTD as defined above.
Measure: Number; unit: Dose Level
Groups:
- Phase I (Stage 1): Stage 1: Patients receive MV-NIS IV over 1 hour on day 1. (Closed to accrual on 12/17/2009 and reopened 10/13/2011)
Arm/Group | Phase I (Stage 1)
Number analyzed (Participants) | 21
Dose Level | 6

3. Primary Outcome: Proportion of Confirmed Response, Defined as a Partial Response (PR) or Better (Phase II)
Description: Confirmed response will be evaluated using all cycles. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 1 year
Population: Only phase II patients who completed the study are included in this analysis. Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating early in Cohort B.
Measure: Number; unit: proportion of patients
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
proportion of patients | 0

4. Secondary Outcome: Overall Toxicity Rate, Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0) (Phase I)
Description: The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below by stage for Phase I patients.
Time Frame: Up to 1 year
Population: Per protocol, Phase I specified secondary endpoint is evaluated for each STAGE independently; thus, the stage 1 dose level groups were combined and the stage 2 dose level groups were combined for this analysis PER PROTOCOL.
Measure: Number; unit: percentage of patients
Groups:
- Phase I: Stage 1 (MV-NIS Alone): Patients receive MV-NIS IV over 1 hour on day 1. (Closed to accrual on 12/17/2009 and reopened 10/13/2011)
- Phase I: Stage 2 (MV-NIS and Cyclophosphamide): Patients receive 10 mg/kg cyclophosphamide IV over 30 minutes and then MV-NIS IV over 1 hour 2 days later. (Temporarily closed to accrual on 10/13/11)
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide)
Number analyzed (Participants) | 21 | 8
percentage of patients | 38 | 25

5. Secondary Outcome: Number of Patients With Clinical Responses (Phase I)
Description: The number of patients with clinical responses (CR, VGPR, PR, or minimal response [MR]) will be summarized by stage.
Time Frame: Up to 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide)
Number analyzed (Participants) | 21 | 8
Participants | 1 | 0

6. Secondary Outcome: Overall Survival (Phase II)
Description: Time from registration to death due to any cause, assessed up to 1 year. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 1 year
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
months | 12.0 [5.6 to NA] — The 95% confidence interval upper limit has not been reached. (insufficient number of participants with events)

7. Secondary Outcome: Time to Progression (TTP) (Phase II)
Description: Time from registration to the earliest date with documentation of disease progression, assessed up to 1 year. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the earliest date with documentation of disease progression, assessed up to 1 year
Population: Phase II specified secondary endpoint will only include Phase II patients. Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating in Cohort B early and to get the overall TTP for Phase II patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
months | 1.48 [1.35 to 240]

8. Secondary Outcome: Progression-free Survival (Phase II)
Description: 1-year progression-free survival (PFS1). Evidence of local recurrence, distant metastasis, or death from any cause within 1 year counted as events in the time-to-event Kaplan-Meier analysis of progression-free survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 1 year
Population: Phase II specified secondary endpoint will only include Phase II patients. Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating early in Cohort B.
Measure: Number; unit: percentage of patients
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
percentage of patients | 6.7

9. Secondary Outcome: Progression-free Survival (Phase II)
Description: 2-year progression-free survival (PFS2). Evidence of local recurrence, distant metastasis, or death from any cause within 2 years counted as events in the time-to-event Kaplan-Meier analysis of progression-free survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 2 years
Population: as for outcome 8
Measure: Number; unit: percentage of patients
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
percentage of patients | 6.7

10. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 5 years
Population: Phase II specified secondary endpoint will only include Phase II patients. Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating in Cohort B early and to get the overall PFS for Phase II patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
months | 1.48 [1.35 to 2.40]

11. Secondary Outcome: Failure-free Survival (Phase II)
Description: Time from registration to the earliest of progressive disease, alternative treatment for myeloma, or death due to any cause, assessed up to 1 year. The distribution of failure-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the earliest of progressive disease, alternative treatment for myeloma, or death due to any cause, assessed up to 1 year
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
months | 1.4783 [1.2155 to 2.3982]

12. Secondary Outcome: Overall Toxicity Rate, Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0) (Phase II)
Description: The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below for Phase II patients.
Time Frame: Up to 1 year
Population: Only phase II patients who completed the study are included in this analysis. Phase II Cohort A and Phase II Cohort B were combined for this analysis due to accrual terminating early in Cohort B and to obtain the overall toxicity rate among Phase II patients.
Measure: Number; unit: percentage of patients
Arm/Group | Phase II (Acetaminophen + Benadryl + MV-NIS)
Number analyzed (Participants) | 15
percentage of patients | 73.3

13. Other Pre Specified Outcome: Time Until Any Treatment Related Toxicity (Phase I)
Description: Tolerability will be explored in an ancillary manner through time-related variables, including time until any treatment related toxicity. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals. The effect of dose and ancillary dichotomized covariates such as age will be explored using log-rank testing involving one covariate at a time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Time Until Hematologic Nadirs (White Blood Cells, ANC, Platelets) (Phase I)
Description: Tolerability will be explored in an ancillary manner through time-related variables, including time until hematologic nadirs. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals. The effect of dose and ancillary dichotomized covariates such as age will be explored using log-rank testing involving one covariate at a time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Time Until Treatment Related Grade 3+ Toxicity (Phase I)
Description: Tolerability will be explored in an ancillary manner through time-related variables, including time until treatment related grade 3+ toxicity. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals. The effect of dose and ancillary dichotomized covariates such as age will be explored using log-rank testing involving one covariate at a time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Biodistribution and Kinetics of Virus Spread
Description: Will be correlated with tumor distribution. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g. Pearson's and Spearman's rho).
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: NIS Gene Expression in Vivo
Description: as for outcome 16
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Radiation Dose
Description: The radiation dose that could be delivered to the bone marrow as well as critical organs such as the liver, lungs and kidneys if iodine-131 were to be administered using MIRDOSE 3 program will be estimated. Where patterns of correlation are indicated, ordinary and partial correlation coefficients (controlling for dose levels) will be calculated. Inferential testing for significant shifts in the correlative laboratory data results across dose levels will be carried out only as a hypothesis generating exercise.
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Viral Replication
Description: Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g. Pearson's and Spearman's rho).
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Viral Shedding
Description: as for outcome 19
Time Frame: Up to 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Only patients who received at least 1 cycle of treatment and submitted AE data are summarized below. Each CTCAE term is a specific event used for medical documentation & is a single MedDRA Lowest Level Term (LLT). Serious AE (SAE) reports may include any serious or non-serious events considered related to the primary event; collectively, these events are referred to as Expedited AEs, & appear in the SAE table. Phase II Cohort A and B combined as they received the same treatment.
Arm/Group | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3 | Phase II (Acetaminophen + Benadryl + MV-NIS)
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 2/4 | 3/4 | 5/7 | 2/3 | 3/3 | 1/2 | 6/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 1/4 | 1/4 | 1/7 | 0/3 | 0/3 | 0/2 | 1/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/4 | 4/4 | 7/7 | 3/3 | 3/3 | 2/2 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 (N=4) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 (N=4) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 (N=7) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 (N=3) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 (N=3) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3 (N=2) | Phase II (Acetaminophen + Benadryl + MV-NIS) (N=15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 1 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 2 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 3 (N=3) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 4 (N=4) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 5 (N=4) | Phase I: Stage 1 (MV-NIS Alone) Dose Level 6 (N=7) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 1 (N=3) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 2 (N=3) | Phase I: Stage 2 (MV-NIS and Cyclophosphamide) Dose Level 3 (N=2) | Phase II (Acetaminophen + Benadryl + MV-NIS) (N=15)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (8) | 3 (10) | 3 (7) | 3 (4) | 4 (7) | 7 (13) | 3 (12) | 3 (10) | 2 (8) | 15 (23)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 10 (11)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (2) | 1 (1) | 3 (5) | 5 (5) | 2 (2) | 3 (4) | 2 (4) | 12 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 8 (9)
Chills (General disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 11 (12)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 13 (13)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 3 (4) | 2 (6) | 1 (1) | 2 (3) | 3 (7) | 1 (1) | 2 (4) | 1 (2) | 1 (4) | 7 (11)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (4) | 3 (5) | 3 (5) | 3 (4) | 3 (4) | 7 (8) | 2 (3) | 3 (6) | 2 (8) | 11 (11)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 2 (4) | 2 (2) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (4) | 3 (6) | 3 (5) | 1 (1) | 3 (4) | 6 (10) | 3 (4) | 2 (5) | 2 (6) | 9 (12)
Platelet count decreased (Investigations) | 3 (8) | 3 (9) | 3 (6) | 1 (1) | 4 (7) | 7 (7) | 3 (6) | 3 (10) | 2 (8) | 13 (13)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (5) | 1 (1) | 2 (3) | 2 (4) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT00450814/Prot_SAP_000.pdf